CLINICAL TRIAL: NCT02926495
Title: Subcutaneous Median Nerve Neuromodulation For Drug-Treatment Resistant Hypertension.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped before start because the project was not fully-funded.
Sponsor: Valencia Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: G160188
Record Dates: First submitted 2016-10-03; First posted 2016-10-06 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Resistant Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Treatment (ON) (Active Comparator)
  Interventions: Device: eCoin System
- Control (OFF) (Sham Comparator)
  Interventions: Device: eCoin System

INTERVENTIONS:
Device: eCoin System — Median nerve neurostimulator.

SUMMARY:
Hypertension is a serious public health issue, affecting approximately 30% of adults. Hypertension greatly contributes to the risk for heart disease and stroke, both among the top three leading causes of death in the Americas, Europe, and Asia. While most treated individuals with hypertension are controlled on medication, diet and exercise, an estimated 12% are resistant to conventional medical intervention. Alternative effective treatments are still needed for this hypertensive patient population to mitigate the risk and incidence of mortality and morbidity.

This original Investigational Device Application is for a study intended to confirm the safety and efficacy of bilateral subcutaneous median nerve stimulation using the eCoin system to treat resistant hypertension. The eCoin device delivers electrical stimulation pulses to the median nerve from a small coin sized device placed under the skin of the distal anterior forearm. The implant delivers a weekly 30 minute treatment based on previous studies showing a long lasting and cumulative effect. The safety and efficacy of eCoin therapy has previously been demonstrated in a multinational, randomized, double-blind, sham-controlled study in New Zealand, Taiwan and Canada.

This trial is a multi-center, prospective, double-blind, 1:1 randomized sham-controlled study of the safety and effectiveness of eCoin median nerve neuromodulation in subjects with drug-treatment resistant hypertension. The eCoin neuromodulation device will be implanted subcutaneously in the right and left forearms of patients with uncontrolled hypertension despite treatment with 3 or more antihypertensive agents. After a 4 week implant healing period, subjects will be 1:1 randomized into either a treatment or control group. One half of the subjects have their devices activated (treatment) and the other half undergo a sham activation (control) to maintain participant blinding to their treatment allocation. During the six months post-randomization, the eCoin is ON in the treatment group and OFF in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Individual is ≥30 and <75 years of age at the time of randomization.
* Individual is receiving a stable medication regimen including maximally tolerated doses of 3 or more anti-hypertensive medications of different classes, of which one must be a diuretic (with no changes for a minimum of 4 weeks prior to screening) that is expected to be maintained without changes for at least 6 months post randomization.
* Individual has an office systolic BP ≥140 mmHg and ≤180 mmHg and diastolic BP ≥80 mmHg and ≤110 mmHg measured at an initial screening visit and a confirmatory baseline visit.
* Individual has a 24 hour ambulatory systolic BP of ≥135 mmHg and ≤175 mmHg at baseline.

Exclusion Criteria:

* Individual in whom medications are expected to change in the next 9 months (6 months post randomization).
* Individual does not agree to have all study procedures performed, and is not competent and willing to provide written, informed consent to participate in this clinical study.
* Individual has type 1 diabetes mellitus or type 2 diabetes mellitus with an A1C ≥ 9%.
* Individual has experienced, within one year of the screening visit, a myocardial infarction, hospitalized unstable angina pectoris, hospitalized heart failure, TIA or a cerebrovascular accident.
* Individual has a scheduled or planned surgery, cardiovascular intervention, or dialysis in the next six months.
* Individual has hemodynamically significant valvular heart disease for which reduction of BP would be considered hazardous.
* Individual has any serious medical condition with a prognosis of <2 years.
* Individual has significant anemia (hemoglobin <100g/L), thrombocytopenia (platelets <100x10(9) /L) or a severe bleeding disorder eg. hemophilia.
* Individual has known secondary hypertension including primary aldosteronism (other than associated with obstructive sleep apnea).
* Individual has pulmonary hypertension.
* Individual requires chronic oxygen support or mechanical ventilation (e.g., tracheostomy, CPAP, BiPAP) other than nocturnal respiratory support for sleep apnea.
* Individual is pregnant, nursing or planning to become pregnant.
* Individual has known or suspected history of medication non-compliance.
* Individual has known unresolved history of drug use or alcohol dependency, lacks the ability to comprehend or follow instructions, or would be unlikely or unable to comply with study follow-up requirements.
* Individual has undergone renal denervation or baroreflex activation therapy.
* Individual has an estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2.
* Individual has another implantable stimulation device including a cardiac pacemaker, ICD, spinal cord stimulator, brain stimulator, vagus nerve stimulator, peripheral nerve stimulator, or cochlear implant.
* Individual is scheduled to have an MRI.
* Individual is currently enrolled in another investigational drug or device trial that has not reached its primary endpoint.
* Individual is working nights or is on a rotating work schedule.
* Individual has an arm circumference too large or small to allow accurate blood pressure measurement with available devices.
* Individual has a history of carpal tunnel syndrome/wrist surgery or other pre-existing compression or non-compression neuropathy in the forearm, wrist or hands that is incompatible with device placement.

Ages: 30 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11 (Estimated); Primary Completion 2018-05 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Difference in Change in 24-hr SBP Between Groups at 6 Months | From baseline to 6 months post-randomization.
  The difference in 24-hour ambulatory systolic blood pressure change from baseline to 6 months post-randomization between the eCoin neuromodulation ON (Treatment) and eCoin neuromodulation OFF (Control) groups.